CLINICAL TRIAL: NCT02146534
Title: Prolonged-release Fampridine as Adjunct Therapy to Active Motor Training in MS Patients: a Phase IV, Double-blind, Placebo-controlled Study.
Brief Title: Prolonged-release Fampridine as Adjunct Therapy to Active Motor Training in MS Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinique Neuro-Outaouais (Other)
Collaborators: CogState Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAN-FMP-13-10507
Record Dates: First submitted 2014-04-23; First posted 2014-05-26 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fampridine (Experimental): extended release fampridine 10mg BID PO for 14 weeks
  Interventions: Drug: extended release fampridine
- placebo (Placebo Comparator): placebo pill BID PO for 14 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: extended release fampridine — pts will receive Fampyra 10 mg BID PO for the duration of the study
  Other Names: Fampyra
  Arms: fampridine
Drug: Placebo — placebo will be taken PO BID
  Arms: placebo

SUMMARY:
Phase 4, single center, double-blind, placebo-controlled study. Fifty (50) patients with MacDonald criteria (2005) multiple sclerosis will undergo active motor training as per the NeuroGym protocol, consisting of 3 sessions of 1 hour per week for a period of 6 weeks (total of 18 sessions).

Half of the patients will be randomized to receive prolonged-release fampridine 10 mg BID as per label, and the other half will receive a placebo BID.

All patients will continue to take their medication (fampridine or placebo) during a subsequent observational period of 8 weeks. Patients will be evaluated at times -4, 0, 6 and 14 weeks.

Study Objectives:

Primary: To demonstrate that MS subjects treated with prolonged-release fampridine 10mg BID will show greater benefit from active motor training as compared with subjects treated with placebo in terms of incidence of responders, degree of response, and duration of response.

Secondary: To demonstrate that MS subjects treated with prolonged-release fampridine 10mg BID will show greater benefit from active motor training as compared with subjects treated with placebo in terms of quality of life measures.

DETAILED DESCRIPTION:
Rationale for the study

Prolonged-release fampridine (4-aminopyridine) is a voltage-gated potassium channel blocking agent. It relieves conduction block in demyelinated nerve fibers by blocking voltage-gated potassium channels on the paranodal axon membranes in vitro. It enhances synaptic transmission by blocking repolarizing potassium currents thus increasing the size of the presynaptic action potential and thus increasing transmitter release. It has been shown in multiple sclerosis patients to improve walking capabilities as measured by the timed 25 feet walk test by more than 20% in approximately 34% of subjects. Prolonged-release fampridine also has measurable effects on motor evoked potentials with transcranial magnetic stimulation in patients with multiple sclerosis and partial spinal cord injuries.

The brain is a dynamic plastic organ that continuously adapts to the demands made upon it. Prolonged-release fampridine by improving nerve conduction in multiple sclerosis patients has the potential to enhance brain plasticity. Activities or processes that call upon such plasticity could therefore also benefit from prolonged-release fampridine. Active motor training when combined with prolonged-release fampridine in patients with multiple sclerosis could therefore show a larger and more sustained measurable clinical benefit than with active motor training alone.

Prolonged-release fampridine by enhancing brain plasticity through improved nerve conduction in the central nervous system can potentiate the clinical benefits of active motor training as measured via assessments of walking capabilities and quality of life in subjects with multiple sclerosis of varying severity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of McDonald criteria MS of all types and of age 18 and older.
* Subjects who meet the prescribing criteria for Fampyra as per product monograph.
* Therapeutic stability (MS and symptomatic treatment) for 3 months prior to screening and for the duration of the study.
* Pyramidal system functional assessment score of 2 or greater and the ability to complete all the assessments with or without aids.
* Female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment.

Exclusion Criteria:

* Any contraindication to receiving fampridine as per product monograph including but not limited to prior history of epilepsy, renal dysfunction (abnormal serum creatinine), concomitant treatment with cimetidine or quinidine.
* Ongoing treatment with fampridine or prior history of fampridine intolerance or ineffectiveness
* Any other condition that would preclude them from undergoing the NeuroGym training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
change in mobility | over 6 and 14 weeks
  timed 8 minutes walk (T8MW) 6 minutes walk (6MW) five times sit to stand test (FTSST)

SECONDARY OUTCOMES:
change in quality of life | over 6 and 14 weeks
  multiple sclerosis impact scale (MSIS-29) short form health survey (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Francois H Jacques, MD FRCP, Principal Investigator — Clinique Neuro-Outaouais
Locations (1):
- Clinique Neuro-Outaouais, Gatineau, Quebec, Canada

REFERENCES:
- [Derived] Jacques F, Schembri A, Nativ A, Paquette C, Kalinowski P. Prolonged-Release Fampridine as Adjunct Therapy to Active Motor Training in MS Patients: A Pilot, Double-Blind, Randomized, Placebo-Controlled Study. Mult Scler J Exp Transl Clin. 2018 Mar 9;4(1):2055217318761168. doi: 10.1177/2055217318761168. eCollection 2018 Jan-Mar. PMID 29552356